CLINICAL TRIAL: NCT00868829
Title: Firebird2 Cobalt-Chromium Alloyed Sirolimus-Eluting Stent Registry Trial
Acronym: FOCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Junbo Ge, Zhongshan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPMFB22009
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Heart Disease
Keywords: Stent; FireBird2; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Firebird2 (Experimental)
  Interventions: Device: Firebird2

INTERVENTIONS:
Device: Firebird2 — For the patient participated, only Firebird2 Stent will be implanted.
  Other Names: Firebird2 Cobalt-Chromium Alloyed Sirolimus-Eluting Stent

SUMMARY:
The experimental design is a multi-center, prospective, non-controlled, non-randomized, single-arm clinical registry trial. The study will enroll 5,000 patients who receive the Firebird2TM Cobalt-ChromiumAlloyed Sirolimus-Eluting Stent implantation. For patient with multivessel disease, only Firebird 2TM Stent will be implanted. The enrollment of patients will take about 4 months. Clinical follow-up will be at 30 day, 6 month, 12 month, 24 month and 36 month. Patients withdrawing the study due to any reasons will not be replaced.

DETAILED DESCRIPTION:
[Definition and management of adverse event] Adverse event refers to any undesirable clinical event. It may be caused by devices, rapamycin, procedure related complications, or the adjunctive medications (such as aspirin, clopidogrel, ticlopidine, or other anti-platelet agent) used in this study. Self report of adverse events by patients should be encouraged. Patients have a right to inquire any information on adverse event at any time of the study. If an adverse event is confirmed, the investigator should collect all related information and complete the Adverse Event Form.

[Classification of adverse events severity] Mild: Mild adverse event refers to clinical event not interfering patient's daily activities.

Moderate: Moderate adverse event refers to clinical event affecting patient's daily activities.

Serious: Serious adverse event refers to clinical event results in patient's inability to undertake daily activity.

[Management of adverse event] All adverse events occurring during the study period should be documented on Adverse Event Forms. Investigators should provide appropriate treatment for all adverse events and follow up the patient until symptom(s) disappear or remain stable

[Documents Recordkeeping] All CRFs and their other original supporting files (such as the informed consent, the lab report, the process records, medical history, the results of physical examinations and diagnosis, the diagnosis, procedure dates and the records regarding equipment management) must be set up in a secure central location by a research site staff and maintained for at least 2 years upon the notification on the termination or completion of the trial issued by MicroPort Medical.

In case the person in charge of keeping these files cannot keep the trial records continuously due to retirement, transferring or any other reason, the recordkeeping should be handed over to another person who is able to accept this task, and a written notification with the successor's name and address should be sent to MicroPort and the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧18 years
2. Patient being suitable candidate for the implantation of drug-eluting stent at physician's discretion
3. Patient with multivessel disease who receive only Firebird2 Stent
4. Patient agrees to provide informed consent to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures.

Exclusion Criteria:

1. Patient not being suitable candidate for the implantation of drug-eluting stent at physician's discretion
2. Patient with multivessel disease who receive other type of stents instead of only Firebird2 Stent
3. Patient who receive other PCI interventions, such as rotablation, directional coronary atherectomy (DCA), TEC, CRA, laser angioplasty, etc.), in addition to PTCA and stenting
4. Patient refuses to provide informed consent
5. Patient who are not able to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
rate of major adverse cardiac events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang F, Yang J, Qian J, Ge L, Zhou J, Ge J; FOCUS registry investigators. Long-term performance of the second-generation cobalt-chromium sirolimus-eluting stents in real-world clinical practice: 3-year clinical outcomes from the prospective multicenter FOCUS registry. J Thorac Dis. 2016 Jul;8(7):1601-10. doi: 10.21037/jtd.2016.05.11. PMID 27499948